CLINICAL TRIAL: NCT06131073
Title: Effects of Speed Endurance Training on Agility and Functional Performance in Soccer Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0445
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Sports Physical Therapy
Keywords: runner; endurance training

STUDY DESIGN:
Intervention Model Description: Randomized Clinical trial
Who Masked: Outcomes Assessor
Masking Description: assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- speed endurance production (SEP) training along with conventional training. (Experimental): Group A along with conventional regime will be given SEP. It will be given 3 days/week.
  The SEP protocol consisted of 6-8 reps of 20-s all-out bouts interspersed with 120 seconds of passive recovery between repetitions. During each 20-s bout, players carried out single shuttle runs of approximately 140-150 m (70-75 + 70-75 m, depending on the group) at their full maximal effort. SEP protocol will be given 3 times/ week for 8th weeks
  Interventions: Other: speed endurance production (SEP) training along with conventional training.
- conventional exercise (Experimental): * A standardized 10-minute warm-up consisting of jogging .
  * Multidirectional dynamic stretching of lower extremity muscles (Hamstring, Quadriceps Calf), for 30 seconds each
  * Jumping (submaximal ankle and squat jumps) will be used for all soccer players before regime starts
  * Exercises including squats; Nordic hamstrings; core rotations and barbell rowing, lunges , hamstrings kicks, side way lunges, standing chest press, crunches (90s rest); core rotations; bounding jumps and fast shifting lunges Each exercise will consists of 3*10, after each exercise 90 seconds rest will be given. These exercises will be given to 3 times a week for 8 weeks
  Interventions: Other: conventional training

INTERVENTIONS:
Other: speed endurance production (SEP) training along with conventional training. — this include speed endurance training for 3 days in a week for 8 weeks.
  Arms: speed endurance production (SEP) training along with conventional training.
Other: conventional training — this include conventional training for 3 days in a week for 8 weeks.
  Arms: conventional exercise

SUMMARY:
Ethical approval is taken from ethical committee of Riphah International university Randomized Control Trial (RCT) will be conducted at Pakistan Cricket Board (PCB) Lahore, through convenience sampling technique on 44 athletes of soccer which will be allocated using random sampling through computerized generated number into Group A and Group B, 6 athletes will be in each group. Group A (interventional) will be given conventional training along with Speed Endurance Production (SEP) Training. Group B (Control) will be will be given conventional training

DETAILED DESCRIPTION:
A Randomized Control Trial (RCT) will be conducted at Pakistan Cricket Board (PCB) Lahore, through convenience sampling technique on 44 athletes of soccer which will be allocated using random sampling through computerized generated number into Group A and Group B, 6 athletes will be in each group. Group A (interventional) will be given conventional training along with Speed Endurance Production (SEP) Training. Group B (Control) will be will be given conventional training There will be 3 sessions in a week for 8th week. Outcome measures will be agility T-Test to measure agility, speed endurance will be measured by 40 meters sprint test and functional performance will be measured by Yo-Yo Intermittent Recovery Test Level 2. The baseline scoring will be on 1st day, follow up will be taken at 4th week and 8th week. Data will be analyzed during SPSS software version 25. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* • Male Soccer Players will be included

  * Age from 15 to 30 years will be included
  * Soccer athletes that playing from past 6 month to one year will be included

Exclusion Criteria:

* Age above 30 years will be excluded

  * Soccer player with injuries (eg: Ankle sprain, meniscal injury, Hamstring strain) will be excluded
  * Any long-term injury (eg: fracture of lower extremity bones) will be excluded

Ages: 15 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — male
Enrollment: 44 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
agility | pre and 8 weeks post interventional
  agility T-Test to measure agility
speed endurance | pre and 8 weeks post interventional
  will be measured by 40 meters sprint test
functional performance | pre and 8 weeks post interventional
  will be measured by Yo-Yo Intermittent Recovery Test Level

CONTACTS AND LOCATIONS:
Overall Officials: rehan khalid, DPT, Principal Investigator — study principal investigator
Locations (1):
- Pakistan Sport Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pojskic H, Aslin E, Krolo A, Jukic I, Uljevic O, Spasic M, Sekulic D. Importance of Reactive Agility and Change of Direction Speed in Differentiating Performance Levels in Junior Soccer Players: Reliability and Validity of Newly Developed Soccer-Specific Tests. Front Physiol. 2018 May 15;9:506. doi: 10.3389/fphys.2018.00506. eCollection 2018. PMID 29867552
- [Background] Iaia FM, Bangsbo J. Speed endurance training is a powerful stimulus for physiological adaptations and performance improvements of athletes. Scand J Med Sci Sports. 2010 Oct;20 Suppl 2:11-23. doi: 10.1111/j.1600-0838.2010.01193.x. PMID 20840558
- [Background] McCormick A, Meijen C, Marcora S. Psychological Determinants of Whole-Body Endurance Performance. Sports Med. 2015 Jul;45(7):997-1015. doi: 10.1007/s40279-015-0319-6. PMID 25771784
- [Background] Iaia FM, Fiorenza M, Perri E, Alberti G, Millet GP, Bangsbo J. The Effect of Two Speed Endurance Training Regimes on Performance of Soccer Players. PLoS One. 2015 Sep 22;10(9):e0138096. doi: 10.1371/journal.pone.0138096. eCollection 2015. PMID 26394225
- [Background] Skovgaard C, Christiansen D, Christensen PM, Almquist NW, Thomassen M, Bangsbo J. Effect of speed endurance training and reduced training volume on running economy and single muscle fiber adaptations in trained runners. Physiol Rep. 2018 Feb;6(3):e13601. doi: 10.14814/phy2.13601. PMID 29417745